CLINICAL TRIAL: NCT01765907
Title: Antalgic Treatment of Painful Bone Metastases by US-guided High Intensity Focused Ultrasound (HIFU).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theraclion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HIFU/F/BM/Feb2012.
Record Dates: First submitted 2013-01-09; First posted 2013-01-10 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Bone Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIFU (Experimental)
  Interventions: Device: HIFU

INTERVENTIONS:
Device: HIFU

SUMMARY:
Antalgic treatment of painful bone metastases by US-guided High Intensity Focused Ultrasound (HIFU).

DETAILED DESCRIPTION:
Inclusion Criteria

* 18 years of age or older.
* Histologically proven malignancy of primary tumor. Histologic diagnosis may be established from needle biopsy, cytology, or a surgical biopsy or resection. If the nature of the lesion has been previously through biopsy, the lesion to be treated does not require further documentation.
* Metastatic disease documented either by imaging techniques (plain radiographs, radionuclide bone scans, computed tomography scans and magnetic resonance imaging) or by histology. Other imaging techniques may be acceptable with the approval of the principal investigator.
* ≤ 3 treatable painful bone metastases.
* "Worst Pain Score" of > 3 on a scale of 10 during a 24-hour period (as scored on the Brief Pain Inventory [BPI] question #3: 0 = no pain; 10 = worst possible pain) despite level II analgesic medications.
* Prothrombin time (PT) >50%, Thrombocytes >50x109/L.
* Estimated life expectancy of 3 months or greater, as estimated by the responsible clinician.
* Targeted tumor clearly visible in B-mode ultrasonography, and accessible to US-HIFU treatment, based on imaging data.
* Agreement from the anaesthetist for a IV conscious sedation
* Signed study-specific informed consent prior to inclusion.
* Negative pregnancy test before inclusion for women of childbearing and or efficient method of contraception.
* Patient with social security coverage. Biphosphonate, chemotherapy or hormone therapy intake should remain stable (if possible) throughout follow-up duration.

Exclusion criteria for subject selection

* Pregnant or lactating women.
* Radiation therapy to the targeted sites within 30 days prior to enrollment.
* Targeted tumor mass is less than 10 mm from spinal cord, nerve bundles, bladder, bowel, or hollow viscera,
* Targeted tumor located in skull (including facial bones), vertebral body or sternum.
* Site at need for surgical stabilization
* Uncontrolled bleeding disorders.
* Hematologic primary malignancies.
* patient participating in other trials using drugs or devices

ELIGIBILITY:
Inclusion Criteria:

* • 18 years of age or older.

  * Histologically proven malignancy of primary tumor. Histologic diagnosis may be established from needle biopsy, cytology, or a surgical biopsy or resection. If the nature of the lesion has been previously through biopsy, the lesion to be treated does not require further documentation.
  * Metastatic disease documented either by imaging techniques (plain radiographs, radionuclide bone scans, computed tomography scans and magnetic resonance imaging) or by histology. Other imaging techniques may be acceptable with the approval of the principal investigator.
  * ≤ 3 treatable painful bone metastases.
  * "Worst Pain Score" of > 3 on a scale of 10 during a 24-hour period (as scored on the Brief Pain Inventory [BPI] question #3: 0 = no pain; 10 = worst possible pain) despite level II analgesic medications.
  * Prothrombin time (PT) >50%, Thrombocytes >50x109/L.
  * Estimated life expectancy of 3 months or greater, as estimated by the responsible clinician.
  * Targeted tumor clearly visible in B-mode ultrasonography, and accessible to US-HIFU treatment, based on imaging data.
  * Agreement from the anaesthetist for a IV conscious sedation
  * Signed study-specific informed consent prior to inclusion.
  * Negative pregnancy test before inclusion for women of childbearing and or efficient method of contraception.
  * Patient with social security coverage.

Exclusion Criteria:

* • Pregnant or lactating women.

  * Radiation therapy to the targeted sites within 30 days prior to enrollment.
  * Targeted tumor mass is less than 10 mm from spinal cord, nerve bundles, bladder, bowel, or hollow viscera,
  * Targeted tumor located in skull (including facial bones), vertebral body or sternum.
  * Site at need for surgical stabilization
  * Uncontrolled bleeding disorders.
  * Hematologic primary malignancies.
  * patient participating in other trials using drugs or devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To assess safety including adverse and serious adverse events, local and systemic tolerance of HIFU in patients with bone metastasis acoording to the Common Terminology Criteria for Adverse events (CTCAE version 4.3) | up to 3 months after HIFU session

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Gustave Roussy, Villejuif, France